PRINCIPAL INVESTIGATOR: Charalampos Floudas, MD, DMSc, MS

STUDY TITLE: Phase I/II Trial of HPV Vaccine PRGN-2009 Alone or in Combination with

Anti-PD-L1/TGF-β trap (M7824) in Subjects with HPV Associated Cancers

**STUDY SITE:** NIH Clinical Center

Cohort: *Phase II Participants*Consent Version: 04/25/2023

## WHO DO YOU CONTACT ABOUT THIS STUDY?

Principal Investigator: Charalampos Floudas, MD, DMSc, MS

Phone: 240-858-3032

Email: charalampos.floudas@nih.gov

## KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you in making your decision about participating in this study. Additional information that may help you make a decision can be found in other sections of the document. Taking part in research at the NIH is your choice.

This study consists of 2 phases.

You are being asked to take part in the Phase II part of the study because you have been newly diagnosed with stage I (T1,2 N1)/II/III p16-positive oropharyngeal cancer or with operable stage II/III/IVA/IVB HPV+ sinonasal squamous cell cancer.

The purpose of Phase II part of research study is to determine if HPV vaccine is able to cause a better immune response after treatment when compared with pre-treatment. The time-period between your cancer diagnosis and standard therapy gives us an opportunity to test these immunotherapy drugs. We also want to find out if giving you immunotherapy before standard therapy helps prevent your tumor from coming back in the future.

The study drug you will receive is called immunotherapy:

• HPV vaccine (PRGN-2009) is a type of vaccine which is designed to teach your immune system how to target and kill cancer cells.

The use of HPV vaccine in this study is considered investigational, which means that this drug has not been approved by the U.S. Food and Drug Administration (FDA) to treat HPV associated cancers. However, the FDA has given us permission to use the HPV vaccine in this study.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Version Date: 04/25/2023


Whether you choose to take part in this study or not, your cancer treatment given by your regular cancer doctors will not change. This study adds the use of this immunotherapy drug (HPV vaccine) before the treatment you will receive as part of your standard cancer treatment for your oropharyngeal cancer.

Side effects can occur with immunotherapy drugs as explained later in the consent. By participating in this study, you will be at risk of experiencing these side effects.

You will have treatment with an HPV vaccine, PRGN-2009. A safe dose of the HPV vaccine has been decided based on Phase I part of the study.

If you decide to join this study, here are some of the most important things that you should know that will happen:

- Once you meet the study requirements to enroll in Phase II, you will receive the immunotherapy drug as follows:
  - o HPV vaccine will be given by injection under the skin on Day 1 and Day 15.
  - You will return 1-2 weeks after the second dose for additional research blood work, imaging, and tumor biopsy.
  - You will then be sent back to your regular cancer doctor for standard therapy and any required treatment such as radiation after your standard therapy. The standard treatment is not part of this Phase II study.
- Each treatment will be given in the Oncology Outpatient Center and will take approximately 2-4 hours.
- You will be seen regularly during the study. You will have clinical, laboratory, and imaging tests to see how you are doing and to see if your disease is responding to the treatment. We will also collect required samples from you (such as saliva, blood and tumor biopsies) for both clinical and research purposes.
- About four weeks after your study therapy has ended, you will be seen in the clinic and possibly have more labs. These visits are important for your safety and if you cannot come to the NIH in person, you will be contacted by phone for follow-up.
- We will contact you for long term follow-up every year, for 5 years after your surgery or chemoradiotherapy, to ask about any adverse events, further treatment of your tumor, and your survival.
- You may experience side effects from taking part in this study. Some can be mild or very serious, temporary, long-lasting, or permanent, and may include death. Examples of some of the side effects include:
  - o Fatigue
  - o Fever
  - o Headache
  - Muscle aches
  - o Injection site reaction

A more complete list of possible side effects is described later in this consent. It is important that you read and understand the possible risks.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


Just as we do not know what side effects you might have, we cannot know if you may benefit from taking part in this study. If you do not benefit, this study and the results from our research may help others in the future.

You are free to stop participating in the trial at any time. If you decide to stop, the study doctor may ask you to agree to certain tests to make sure it is safe for you to stop.

The remaining document will now describe more about the research study. This information should be considered before you make your choice. Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research interventions in which they would want to participate. Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

If the individual being asked to participate in this research study is not able to give consent to be in this study, you are being asked to give permission for this person as their decision-maker. The term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research, throughout the remainder of this document.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

This study has two phases.

The purpose of the Phase II part of this research study is to determine if the HPV vaccine is able to result in a better immune response post-treatment when compared with pre-treatment. We also want to find out if giving you immunotherapy before standard therapy helps prevent your tumor from coming back in the future.

You are being asked to take part in the Phase II part of the study because you have been newlydiagnosed with stage II or III p16-positive oropharyngeal cancers.

The use of HPV vaccine in this study is considered investigational, which means that this HPV vaccine has not been approved by the U.S. Food and Drug Administration (FDA) to treat HPV associated cancers. However, the FDA has given us permission to use the HPV vaccine in this study.

#### WHAT WILL HAPPEN DURING THE STUDY?

Below is a description of what will be asked of you and what will occur if you decide to take part in this study.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




# Before you begin the study

To determine if you can be a part of this study, you will need to have the following tests and procedures. These may be done under a separate protocol:

- Medical history and physical examination including height, weight, and vital signs;
- CT scan of the neck and chest (if you have oropharyngeal cancer or sinonasal squamous carcinoma);
- CT scan of the skull (only if you have sinonasal squamous carcinoma);
- Routine blood tests;
- EKG;
- For skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion;
- Pregnancy test for women who are able to have children;
- Hepatitis B and C screening tests;
- HIV screening test;
  - As part of this study, we will test you for infection with HIV, the virus that causes AIDS. If you are infected with HIV, you may still be able to take part in this study. We will tell you what the results mean, how to find care, how to avoid infecting others, how we report HIV infections, and the importance of informing your partners at possible risk because of your HIV infection.
- Urine tests;
- Confirmation of your disease. If there is no available tumor sample or pathology report, a biopsy will be performed to confirm the diagnosis.

## **During the study**

Once we know that you are eligible and you sign the consent document agreeing to participate in the study, you may need to have some of the tests that were done at screening repeated depending on how much time has passed. Your study team will let you know if any of the following tests need to be repeated on Week 1 Day 1.

- Medical history and physical examination including height, weight, and vital signs;
- CT scan of the neck and chest and/or MRI;
- CT scan of the skull and/or MRI (only if you have sinonasal squamous carcinoma);
- Routine blood and urine tests;
- Pregnancy test for women who are able to have children (within 5 days before starting drug treatment);
- Hepatitis B and C screening tests;
- HIV screening test;
- EKG to check your heart;
- Assessment of hypersensitity, if required;
- For skin lesions: color photography, if needed;
- Tumor markers.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


During your participation you will receive the HPV vaccine as explained in Key Information section above.

• You will receive the HPV vaccine by injection under the skin on Day 1 and Day 15.

We will continue to take assessments, such as physical exam, weight, vital signs, EKG, collection of blood for routine lab testing, tumor markers, pregnancy test for women of childbearing age, and scans for the evaluation of your tumor, during your participation.

# Additional research testing

In addition to the tests that we will conduct to determine whether you are having side effects or if you are responding to the study therapy, we will also collect samples from you for purposes of research only. The samples are being tested to look at the effects of therapy on your immune system and markers of tumor activity, including collecting and testing tumor cells, as well as development of anti-vector antibodies (AVA) in response to the therapy..

The samples for these studies include:

- Blood Tests: When possible, research blood (4-5 tablespoons) will be collected at baseline, and at Weeks 1, 3, and 5.
- Tumor Biopsy: Tissue sample will be collected at Week 1 Day 1 as well as at Week 5 by an ENT doctor under direct visualization. The first biopsy at Week 1 will not need to be done if you had a biopsy done outside of NIH (within the past 6 months) and we can be given a sample of that biopsy.
- Saliva Sample: Depending on the type of cancer you have, we may collect saliva with a mouth rinse several times during the study.

In this study we will perform genetic testing on your RNA. RNA (ribonucleic acid) carries instructions from your DNA (deoxyribonucleic acid) to the parts of the cells that makes proteins. We will perform limited genetic testing on certain immune cells in your blood and tumor samples to characterize changes in the RNA of a particular molecule located on the immune cell. We will perform further genetic testing on your blood samples, looking at how much RNA you have for certain panels genes. This helps us to learn how active the genes are.

# When you are finished with treatment

End of Treatment Visit

If you stop participation in the study before the completion of one year of treatment, then you will be asked to come into the clinic on the day of or within 7 days of the decision to stop treatment for the following tests and procedures: physical examination including weight, and vital signs; EKG; routine blood tests to measure blood chemistry and complete blood count; pregnancy test if you are a woman who can have children; and scans if you stop study therapy before your disease worsens.

Safety Visit

After your treatment ends or if you stop participation in the study for any reason you will be asked to come into the clinic for a 28 day follow-up visit or telephone call following your last dose of study drug(s).

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


During the visit the following tests and procedures will be given: physical examination including weight and vital signs; EKG; and routine blood tests; and pregnancy test if you are a woman who can have children.

Long Term Follow-up

We will also contact you for long term follow-up every year, for 5 years after completion of your surgery or chemoradiotherapy.

If your disease has progressed while being treated then you will be followed by phone or email for any adverse events, further treatment of your tumor, and your survival.

If your disease did not progress while being treated then you will receive tumor scans until progression of your disease and will be followed by phone or email for any adverse events, further treatment of your tumor, and your survival. If you completed one year of treatment on this study then you may be asked to complete an additional year of treatment at the time of your disease progression. After that one year a follow-up visit may be required if determined by your study doctor.

#### HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this study, the treatment portion is expected to last for about one month for Phase II. After the treatment part is completed, we will continue to follow you for 5 years, until the study ends, or you decide to stop participating.

#### HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

We plan to have approximately 22 people participate in the Phase I part of the study and 22 people in the Phase II part of the study at the NIH.

# WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

#### **Risks from Study Therapy**

# Side Effects of HPV Vaccine (PRGN-2009)

This is a first in human study with PRGN-2009. Possible side effects may include injection site reaction, fever, flu like symptoms (e.g., fatigue, headache, muscle aches), poor appetite, increase in blood sugar, and skin rash.

For patients with local cancer, there is a risk of having delays in standard therapy (e.g., surgery or radiation) which may result in a reduced chance of being cured from cancer.

If any of these side effects occur, you must inform your study doctor immediately.

## **Other Risks**

#### Risk from Blood Collection

Risks of blood draws include pain and bruising in the area where the needle is placed, lightheadedness, and rarely, fainting. When large amounts of blood are collected, low red blood cell count (anemia) can develop.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


#### CT Scan Risk

CT scans create low levels of radiation, which has a small potential to cause cancer and other defects. However, the risk associated with one scan is small.

## Risks Due to Contrast Agents for CT

You may receive a contrast agent as part of your CT scan. Contrast agents can cause allergic reactions and kidney damage. Allergic reactions can include mild itching associated with hives but can also result in a serious life-threatening emergency from difficulty breathing. If this occurs, it is treatable.

# Risks of Biopsy Using Clinical Endoscopy and Nasopharyngo-laryngoscopy

In this procedure, a physician gently places a small, thin, flexible endoscope with a camera down through your nose to view your upper airway anatomy above the vocal cords. This procedure takes only a few minutes, is painless and does not require any sedation. It is a normal part of an ENT exam. Risks of clinic endoscopy include bleeding from nose or sudden drop in heart rate if body reacts to certain triggers, each of which occur in <1% of all patients.

If your tumors are not accessible in the clinic or a biopsy in the clinic is deemed unsafe by the study doctor, biopsies may be performed in the operating room under general anesthesia. Side effects of general anesthesia may include temporary confusion, difficulty passing urine, bruising or soreness from the IV drip, nausea and vomiting, shivering and feeling cold, and sore throat. Risks of operative biopsies include post-op bleeding (<1% of all patients), dental damage from laryngoscopy instrumentation (<1% of all patients) and temporary tongue abnormal sensation (<10% of all patients) that resolves within a few days.

## Risk from Saliva Collection

Saliva collection is not known to be associated with risk. You may have some discomfort from the oral rinse and gargle with saline.

#### **MRI**

Magnetic resonance imaging (MRI) uses a strong magnetic field and radio waves to take pictures of the body. If you have a history of metastases to your brain or if we are concerned that you may have metastases to your brain, we will obtain pictures of your brain for this study. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, you will lie on a table that can slide in and out of the cylinder. We will place soft padding or a coil around your head. You will be in the scanner about 30 minutes. You may be asked to lie still for up to 30 minutes at a time. While in the scanner you will hear loud knocking noises, and you will be fitted with earplugs or earmuffs to muffle the sound. You will be able to communicate with the MRI staff at all times during your scan, and you may ask to be moved out of the machine at anytime.

It is very important for the experiment that you do not move your head or body inside the scanner. We will use padding around your head to help keep it in place.

We may place a bar in your mouth to help keep your head still.

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


# Risks for MRI

People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

# Risks of Gadolinium enhanced MRI

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (iv) catheter. It will be done for research and medical purposes.

It is not known if MRI with contrast is completely safe for a developing fetus. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each MRI scan with contrast. The scan will not be done if the pregnancy test is positive.

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis (NSF)". This condition always involves the skin and can also involve the muscles, joints and internal organs. NSF has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is below the safe level.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA has issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Version Date: 04/25/2023




effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain in the body than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain in the body. We will also give you additional information called a "Medication Guide." Upon request, we will give you individual information about retained gadolinium we see on your studies.

# Risks of Delaying Potentially Curative Treatment

Side effects of this investigational treatment may cause delay in your scheduled curative therapy. A prior study has shown that people with oropharyngeal cancer who received treatment more than 10 weeks after their initial diagnosis did significantly worse than those who received treatment sooner.

# What are the risks related to pregnancy?

If you are able to become pregnant, we will ask you to have a pregnancy test before starting this study. You will need to practice an effective form of birth control before starting study treatment, during study treatment, and for 2 months after you finish study treatment (the restricted period).

If you become pregnant, there may be unknown risks to the fetus or unborn child, or risks that we did not anticipate. There may be long-term effects of the treatment being studied that could increase the risk of harm to a fetus. You must tell the study doctor if your birth control method fails during the restricted period. If you think or know you have become pregnant during the restricted period., please contact the study team soon as possible.

If you are a sexually active person with a partner able to become pregnant, it is important that your partner not become pregnant during the restricted period. There may be unknown risks to the fetus or risks we did not anticipate. You and your partner must agree to use birth control if you want to take part in this study. If you think your partner has become pregnant during the restricted period, please contact the study team as soon as possible. If you and your partner plan for your partner to become pregnant after the restricted period, please discuss this with the study team.

## What are the risks of radiation from being in the study?

During your participation in this research study, you will be exposed to radiation from 3 CT scans. The amount of radiation exposure you will receive from these procedures is equal to approximately 0.99 rem or 1.29 rem depening on your type of cancer. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The CT scans that you get in this study will expose you to the roughly the same amount of radiation as 3.3 or 4.3 years' worth of background radiation, depending on your type of cancer. Most of the time, this amount of extra radiation is not harmful to you. However, scientists believe that being exposed to too much radiation can cause harmful side effects. This could include gettinga new cancer. We estimate that this could happen in about 1 out of every 1000 people who get a very large amount of extra radiation.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Version Date: 04/25/2023  You may not participate in this study if you are pregnant. If you are able to become pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

# Protections against misuse of genetic information

This study involves genetic testing on samples. Some genetic information can help predict future health problems of you and your family and this information might be of interest to your employers or insurers. The Genetic Information Nondiscrimination Act (GINA) is a federal law that prohibits plans and health insurers from requesting genetic information or using genetic information. It also prohibits employment discrimination based on your health information. However, GINA does not address discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed condition or disease that has a genetic component.

## WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You might not benefit from being in this study.

However, the potential benefit to you might be a reduction in the size of your tumor which may or may not have favorable impact on symptoms and/or survival.

## Are there any potential benefits to others that might result from the study?

There is a need for new treatments in patients with advanced HPV associated cancers as standard therapies often do not work. In the future, other people might benefit from this study because of the knowledge gained from the outcome of this trial using a novel immunotherapy.

#### WHAT OTHER OPTIONS ARE THERE FOR YOU?

Before you decide whether or not to be in this study, we will discuss other options that are available to you. Instead of being in this study, you could:

- choose to be treated with surgery, radiation or with drugs already approved by the FDA for your disease;
- choose to take part in a different study, if one is available;
- choose not to be treated for cancer but you may want to receive comfort care to relieve symptoms.

You should discuss with your doctor your other choices and their risks and benefits.

#### DISCUSSION OF FINDINGS

#### New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


#### EARLY WITHDRAWAL FROM THE STUDY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest;
- if your disease worsens or comes back during treatment;
- if you have side effects from the treatment that your doctor thinks are too severe;
- if you become pregnant;
- if the HPV vaccine becomes unavailable;
- if new information shows that another treatment would be better for you;
- if you do not follow the study rules;
- if the study is stopped for any reason.

In this case, you will be informed of the reason therapy is being stopped.

After therapy is stopped we would like to see you for a safety visit 28 days after your last dose.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to Precigen, Inc. or designated representatives.

# STORAGE, SHARING AND FUTURE RESEARCH USING YOUR SPECIMENS AND DATA

# Will your Specimens or Data be Saved for Use in Other Research Studies?

As part of this study, we are obtaining specimens and data from you. We will remove all the identifiers, such as your name, date of birth, address, or medical record number and label your specimens and data with a code so that you cannot easily be identified. However, the code will be linked through a key to information that can identify you. We plan to store and use these specimens and data for studies other than the ones described in this consent form that are going on right now, as well as studies that may be conducted in the future. These studies may provide additional information that will be helpful in understanding HPV associated cancers or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or devices, that may lead to the development of a commercial product by the NIH and/or its research or commercial partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you.

| I give permission | for my co | oded spec | imens an | d data to | be store | d and | used for | or future | research | ı as |
|---|---|---|---|---|---|---|---|---|---|---|
| described above. | | | | | | | | | | |

| Yes | No |
|----------|-----------------|
| Initials | <b>Initials</b> |

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) File in Section 4: Protocol Consent (2) Version Date: 04/25/2023


## Will Your Specimens or Data Be Shared for Use in Other Research Studies?

We may share your coded specimens and data with other researchers. If we do, while we will maintain the code key, we will not share it, so the other researchers will not be able to identify you. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or commercial entities.

I give permission for my coded specimens and data to be shared with other researchers and used by these researchers for future research as described above.

| Yes | No |
|----------|----------|
| Initials | Initials |

If you change your mind and do not want us to store and use your specimens and data for future research, you should contact the research team member identified at the top of this document. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your specimens and data. For example, if some research with your specimens and data has already been completed, the information from that research may still be used. Also, for example, if the specimens and data have been shared already with other researchers, it might not be possible to withdraw them.

In addition to the planned use and sharing described above, we might remove all identifiers and codes from your specimens and data and use or share them with other researchers for future research at the NIH or other places. When we or the other researchers access your anonymized data, there will be no way to link the specimens or data back to you. We will not contact you to ask your permission or otherwise inform you before we do this. We might do this even if you answered "no" to the above questions. If we do this, we would not be able to remove your specimens or data to prevent their use in future research studies, even if you asked, because we will not be able to tell which are your specimens or data.

NIH policies require that your clinical and other study data be placed in an internal NIH database that is accessible to other NIH researchers for future research. These researchers will not have access to any of your identifiers, such as your name, date of birth, address, or medical record number; and your data will be labeled with only a code. We cannot offer you a choice of whether your data to be placed in this database or not. If you do not wish to have your data placed in this database, you should not enroll in this study.

# Will Your Genomic Data Be Shared Outside of This Study?

As part of this research study, we will put your genomic data in a large database for broad sharing with the research community. These databases are commonly called data repositories. The information in this database will include but is not limited to genetic information, race and ethnicity and sex. If your individual research data are placed in one of these repositories, they will be labeled with a code and not with your name or other information that could be used to easily identify you, and only qualified researchers will be able to access them. These researchers must receive prior approval from individuals or committees with authority to determine whether these researchers can access the data.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17) File in Section 4:

File in Section 4: Protocol Consent (2) Version Date: 04/25/2023


NIH policies require that genomic data be placed in a repository for sharing. Therefore, we cannot offer you a choice of whether your data will be shared. If you do not wish to have your data placed in a repository, you should not enroll in this study.

# **How Long Will Your Specimens and Data be Stored by the NIH?**

Your specimens and data may be stored by the NIH until they are no longer of scientific value or if you withdraw consent for their continued use, at which time they will be destroyed. Your specimens and data may be stored by the NIH indefinitely.

# Risks of Storage and Sharing of Specimens and Data

When we store your specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity, for example, when appropriate, we remove information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or that no one will gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your specimens and data.

## COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of you participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Version Date: 04/25/2023

Page **13** of **17** 



# **CONFLICT OF INTEREST (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

The NIH and the research team for this study are using:

• HPV vaccine (PRGN-2009) developed by Precigen, Inc.

through a joint study with your study team and this company. This company also provides financial support for this study.

#### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor (Center for Cancer Research) or their agent(s)
- Qualified representatives from Precigen, Inc., the pharmaceutical company who produces HPV vaccine, or their agent(s).

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by the court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA); or
- 3. is for other research; or
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

#### **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical information we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Version Date: 04/25/2023


#### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

## PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Charalampos Floudas, MD, charalampos.floudas@nih.gov, 240-858-3032. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

#### CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Version Date: 04/25/2023




| | I consent to participate in this study. | |
|---|---|---|
| Signature of Research Participant | Print Name of Research Participa | ant Date |
| about this study and have been given to make research decisions on beh | tive (LAR) for an Adult Unable to Consent: wen the opportunity to discuss it and to ask questical of the adult participant unable to consent and hele, the information in the above consent was described in the study. | ons. I am legally authorize ave the authority to prove |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| <u>-</u> | her:<br>ocess has been used to enroll a non-English spo<br>the full consent has been used to enroll a blind | - · |
| <u>-</u> | ocess has been used to enroll a non-English spo | _ • |
| 2. An oral presentation of the signature of Witness NIH ADMINISTRATIVE SE INTERPRETER: An interpreter, or other indiv | ocess has been used to enroll a non-English specific full consent has been used to enroll a blind | Date ING THE USE OF A |
| 2. An oral presentation of the Signature of Witness NIH ADMINISTRATIVE SE INTERPRETER: An interpreter, or other indivities administration of informed coalso serve as the witness. An interpreter, or other indivities and interpreter, or other indivities and interpreter, or other indivities and interpreter. | ocess has been used to enroll a non-English specific full consent has been used to enroll a blind Print Name of Witness CTION TO BE COMPLETED REGARDI idual, who speaks English and the participant's print of | Date Date The USE OF A referred language facilitate obtaining consent may referred language facilitate of the person |


IRB NUMBER: 20C0104 IRB APPROVAL DATE: 4/25/2023